CLINICAL TRIAL: NCT05630170
Title: Pilot Evaluation for SMartphone-adaptable Artificial Intelligence for PRediction and DeTection of Left Ventricular Systolic Dysfunction
Brief Title: The SMART-LV Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2000034006; No NIH funding (Other: 12.08.23)
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: In the ECG repository of Yale New Haven Hospital, all patients undergoing a 12-lead screen in an outpatient setting, from whom 20 individuals, 10 each with high and low predicted probability of LVSD, will be invited for a limited echocardiogram to definitively evaluate for LVSD. The investigators will assess whether the AI-ECG model continues to have the reported discrimination and sensitivity of >90% for LVSD diagnosis in a screening setting in outpatient routine clinical care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-ECG (Experimental): A novel AI-ECG model developed at the Cardiovascular Data Science (CarDS) lab will be used as Software as Medical Device (SaMD) on ECG images for detection of LVSD.The AI-ECG model will be used on all participants undergoing a 12-lead ECG.
  Interventions: Device: AI-ECG

INTERVENTIONS:
Device: AI-ECG — A novel AI-ECG model developed at the Cardiovascular Data Science (CarDS) lab will be used as Software as Medical Device (SaMD) on ECG images for detection of LVSD.

SUMMARY:
The goal of this pilot study is to evaluate the prospective performance of an image-based, smartphone-adaptable artificial intelligence electrocardiogram (AI-ECG) strategy to predict and detect left ventricular systolic dysfunction (LVSD) in a real-world setting.

DETAILED DESCRIPTION:
The SMART-LV pilot study will be a prospective cohort study in outpatient clinics at the Yale New Haven Hospital. Participants who have undergone a 12-lead electrocardiogram (ECGs) with either a high (≥80%) or low (<10%) probability of LVSD on AI-ECG algorithm, but without an echocardiogram done in the clinical setting for at least 90 days after the ECG, will be identified by electronic health record (EHR) and invited for a limited echocardiogram/cardiac ultrasonogram for assessing LV ejection fraction. The goal of the study is to evaluate the feasibility of recruiting patients and performing the study after pursuing a screening on 12-lead ECGs. The procedure currently used for detection of LVSD, echocardiograms, are inaccessible and expensive. Therefore, while AI-ECG-based algorithms using a smartphone- or web-based application can broaden access to screening, a thorough evaluation for this indication is needed before clinical adoption. The investigators intend to use the results as pilot data for sample size and drop-off rate estimation for a subsequent larger prospective cohort study aimed at validating the performance characteristics of the model in a screening setting.

The validation of this accessible ECG-based screening strategy, that can be directly used by clinicians using a smartphone or web-based application, can transform the early identification of LVSD before the development of symptoms, thereby allowing broader utilization of evidence-based therapies to prevent symptomatic heart failure and premature death.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Patients who have undergone a prior echocardiogram.
* Patients with a prior diagnosis of left ventricular dysfunction, based on a documented low ejection fraction (EF) in the medical record.
* Patients with an intermediate predicted probability of low EF (10 to 80%)
* Patients with a prior diagnosis of heart failure as determined by International Classification of Diseases-10 diagnosis code for heart failure.
* Research opt-out patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Successful detection of asymptomatic LVSD by AI-ECG | During study visit approximately 50 minutes
  Device feasibility of AI-ECG will be evaluated by comparing the proportion of patients with LVSD on echocardiography among those with a high predicted probability of LVSD on an AI-ECG screen compared with the proportion of patients with LVSD on echocardiography in those with a negative AI-ECG screen. Higher proportions indicate successful detection of asymptomatic LVSD compared with routine clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Khera, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States